CLINICAL TRIAL: NCT03494283
Title: Prospective Epidemiological Study of Injuries Encountered in the Practice of CrossFit in Grand Nancy Clubs Over a Period of 8 Months.
Brief Title: CrossFit's Injuries Study in Grand Nancy Clubs During 2018-2019
Acronym: CROSSFIT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02825-48
Record Dates: First submitted 2017-12-15; First posted 2018-04-11 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: CrossFit Injuries
Keywords: CrossFit injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CrossFit injuries
  Interventions: Behavioral: Practice Behaviour

INTERVENTIONS:
Behavioral: Practice Behaviour — Improve and modify practice of the practicers and of the professionals who are framing to decrease the injury incidence.

SUMMARY:
CrossFit is a recent sport that has been democratized since the beginning of the 2000's in France. The 3 major studies of CrossFit injuries were conducted in the United States in 2014, Brazil in 2016 and the United States in 2017. They show a discrepancy in terms of injuries average, from 19.4% to 31% in relation to an upsurge in the number of CrossFit practitioners, the specific training or not of the coaches framing this activity, the practice or not in competition. The main locations of these wounds are highlighted at the shoulders, lumbar region and knees. In France, to date, no epidemiological studies have been conducted on this subject.

Hypothesis: High incidence of injuries related to a lack of framing, or bad practice and ignorance of CrossFit practitioners.

Objectives : Estimate the injuries incident due to the CrossFit practice over a 8-month period in an adult population who practice in clubs .

Research, among the anthropometric, sociodemographic, environmental, and the nature and frequency of practice and training sessions, those which are associated with the occurrence of injury in this cohort.

ELIGIBILITY:
Inclusion Criteria:

Men and women

* 18 years and over
* Practicing CrossFit in a club of the Grand Nancy
* Information and non-opposition to research

Exclusion Criteria:

* Opposition to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women
  * 18 years and over
  * Practicing Crossfit in a club of the Grand Nancy
  * Information and non-opposition to research
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
CrossFit's injuries follow-up questionaire | each month during 8 months
  Questionaire about musculoskeletal pain or discomfort due to CrossFit practice during the previous month .For a period of 8 months, in a population of adults practicing in a club, with musculoskeletal injuries questionaire. A questionaire is given each month during 8 months concerning the previous month ( Questions about physical pain that they felt, practice modification... )This questionaire is not validated.

SECONDARY OUTCOMES:
CrossFit's injuries inclusion questionaire . | At inclusion
  One questionaire is given at inclusion for baseline demographic and baseline data (Age, sex , size , work's condition, practiced sports ) . At the end of the study, the goal is to relate these data to the incidence of injuries found .This questionaire is not validated.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Nancy, France

IPD SHARING:
Plan to Share IPD: No